CLINICAL TRIAL: NCT00653237
Title: A Comparison of The Laryngeal Mask Supreme™ and the I-gel™ in a Simulated Difficult Airway Scenario in Anesthetized and Ventilated Patients
Brief Title: Laryngeal Mask Supreme™ Versus the I-gel™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: igellma-1
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Patients Undergoing Elective General Anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): crossover trial. insertion of both devices consecutively, computer randomized order
  Interventions: Device: I-gel and LMA Supreme: supraglottic airway devices

INTERVENTIONS:
Device: I-gel and LMA Supreme: supraglottic airway devices — Insertion of a supraglottic airway device
  Other Names: Laryngeal Mask Supreme, supraglottic airway device

SUMMARY:
We evaluate two new developed airway devices, which provide patent airway during general anesthesia. In 60 patients undergoing elective general anesthesia, we will simulate a difficult airway by using an extrication device collar). We then place consecutively both airway devices in the mouth and check for ease of insertion and time used.

DETAILED DESCRIPTION:
The LMA Supreme™ and the I-gel™ are both new developed supraglottic airway devices to provide patent airways during general anesthesia. So far, prospective randomized controlled trials comparing their performance are not yet published. Both devices can be used in difficult airway situations, pre-hospital and in the hospital. In this prospective, randomized, controlled cross-over trial, we are going to evaluate the performance of both devices in a simulated difficult airway scenario using an extrication collar to limit both mouth opening and neck movement. In a maximum total of 60 patients undergoing elective surgery, we will place both airway devices consecutively and ventilate the patients. First attempt success rate and time to success will be recorded. Secondary outcomes include oropharyngeal pressure leak, ease of gastric catheter insertion, adverse events and side effects. Our hypothesis is that no difference exists between the two devices. Our 0-hypothesis is that there is a difference

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3 patients undergoing elective operation

Exclusion Criteria:

* Not speaking german or refusing to participate
* BMI >35, <50kg
* Planned operation time >4h
* High risk of aspiration
* Cervical spine disease, known difficult airway, mouth opening <20mm
* Upper respiratory tract symptoms in the previous 10 days
* Preoperative sore throat
* Poor dentition with high risk of damage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
first attempt success rate and time to success | during intervention

SECONDARY OUTCOMES:
leak pressure | during intervention

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, M.D., Study Director — Department of Anesthesia, University Hospital Berne, Switzerland
Locations (1):
- University Hospital, Bern, Canton of Bern, Switzerland